CLINICAL TRIAL: NCT03983629
Title: French National Registry of Congenital Dyserythropoietic Anemia
Brief Title: Registry of Congenital Dyserythropoietic Anemia
Acronym: CDA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: OBS-0020
Record Dates: First submitted 2019-06-05; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Congenital Dyserythropoietic Anemia
Keywords: Congenital Dyserythropoietic Anemia; French registry
MeSH Terms: conditions — Anemia, Dyserythropoietic, Congenital | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — serum and bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CDA patients
  Interventions: Other: Collection of data and genetic analysis

INTERVENTIONS:
Other: Collection of data and genetic analysis — Data collected are: History of disease, medical history, family medical history, biological results, Imaging results, disease progression Genetic analysis will be performed with whole genome and whole exome sequencing

SUMMARY:
Congenital dyserythropoietic anemia is a heterogeneous inherited disease. Hyperplasic erythropoiesis is ineffective and associated with morphological abnormalities of some of the erythroblasts that form the basis of cytological classification. The cumulative incidence is not very clear, but varies between countries from 0.08 million in Scandinavia to 2.6 cases/million inhabitants in Italy where it appears to be the most reported.

The common manifestation is moderate chronic congenital anemia. This anaemia is either normocytic or discreetly macrocytic, non-regenerative or inappropriate regarding anaemia, contrasting with signs of hemolysis with moderate unconjugated hyperbilirubinemia. Diagnosis is usually made in the pediatric period, but because of the great heterogeneity, the diagnosis sometimes may be delayed. Splenomegaly and jaundice are mostly present. Secondary hemochromatosis is common in the absence of transfusion due to hyper-intestinal absorption of iron induced by the dyserythropoiesis.

The transmission mode for Type I and II is autosomal recessive, while it is autosomal dominant or sporadic for Type III.

Several clinical questions remain concerning this disease :

* the median survival of patients is not well known, neither the causes of death
* benefit/risk of splenectomy
* iron overload quantification and consequences

The idea is to stablish a French registry of congenital dyserythropoietic anemia in order to help to understand the correlation between phenotype and genotype of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed CDA
* No opposition to the use of health data for research purposes

Exclusion Criteria:

* Patient opposed to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with confirmed CDA
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-02-23 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of mutations | up to three years
  Genetic analysis will be performed with whole genome and whole exome sequencing

SECONDARY OUTCOMES:
Median survival | up to three years
Prevalence of different causes of death | up to three years
Rate of Interferon treatment efficacy | up to three years

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Carpentier, MD, Principal Investigator — GHICL
Locations (1):
- Hôpital Saint-Vincent de Paul, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No